CLINICAL TRIAL: NCT04842123
Title: Electrocardiogram Clinical Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Garmin International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ECG-002
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Atrial fibrillation (AF) (Other): Patients with a known history of AF who are in AF at the time of study screening.
  Interventions: Diagnostic Test: Electrocardiogram
- Normal Sinus Rhythm (SR) (Other): Patients with no known diagnosis of AF or other arrhythmia
  Interventions: Diagnostic Test: Electrocardiogram

INTERVENTIONS:
Diagnostic Test: Electrocardiogram — Simultaneous assessment of the heart rhythm determined from a 12-lead ECG and the Garmin ECG software algorithm heart rhythm classification on single-lead ECG data derived from the wearable device. All participants will record three simultaneous 12-lead and single-lead ECGs.

SUMMARY:
The purpose of the study is to confirm the Garmin ECG (electrocardiogram) software algorithm can detect and classify atrial fibrillation and normal sinus rhythm on single lead ECG data derived from a Garmin wrist-worn, consumer device. The study will also confirm the software's ability to create a Lead I ECG that is clinically equivalent to a reference device. The Garmin ECG software is not a diagnostic system and is intended for informational purposes only.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand, and provide written informed consent;
* Willing and able to participate in the study procedures as described in the consent form;
* Individuals who are 22 years of age and older;
* Able to communicate effectively with and follow instructions from the study staff;
* Have a wrist circumference that fits within the device band; and
* For subjects enrolled into the AF population, subjects must have a known diagnosis of AF and be in AF at the time of screening.

Exclusion Criteria:

* Physical disability that precludes safe and adequate testing;
* Mental impairment resulting in limited ability to cooperate;
* Subjects with a pacemaker or implantable cardioverter-defibrillator (ICD);
* Acute myocardial infarction within 90 days of screening or other cardiovascular disease that, in the opinion of the Investigator, increases the risk to the subject or renders data uninterpretable;
* Acute pulmonary embolism, pulmonary infarction, or deep vein thrombosis within 90 days of screening;
* Stroke or transient ischemic attack within 90 days of screening;
* Subjects taking rhythm control drugs;
* Symptomatic (or active) allergic skin reactions such as eczema, rosacea, impetigo, dermatomyositis, or allergic contact dermatitis on both wrists or over electrode attachment sites, including known allergy or sensitivity to silicone bands primarily used in wrist-worn fitness devices;
* Known sensitivity to medical adhesives, isopropyl alcohol, watch bands, or ECG electrodes;
* A history of abnormal life-threatening rhythms as determined by the Investigator;
* Significant tremor that prevents subject from being able to hold still;
* Women who are pregnant at the time of study participation; and
* Subjects enrolled into the SR population must not have any diagnosis of AF.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Specificity of rhythm classification | 1 Day
  Number of participants with a SR software rhythm classification in agreement with a physician's interpretation of heart rhythm based on gold standard 12-lead ECG
Sensitivity of rhythm classification | 1 Day
  Number of participants with an AF software rhythm classification in agreement with a physician's interpretation of heart rhythm based on gold standard 12-lead ECG

SECONDARY OUTCOMES:
Number of ECGs that pass a visual overlay | Day 1
  Number of participants with software's ability to produce a clinically equivalent waveform in agreement to a gold standard Lead I reference
Difference in R-wave amplitudes between the software and gold standard reference | Day 1
  Number of participants with software's ability to produce a clinically equivalent waveform in agreement to a gold standard Lead I reference

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Hope Research Institute, Phoenix, Arizona
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - HealthEast, Saint Paul, Minnesota
  - Northwell Health North Shore University Hospital, Manhasset, New York
  - Northwell Health Lenox Hill Hospital, New York, New York
  - MedStar Health Cardiac Electrophysiology at Fairfax, Fairfax, Virginia